CLINICAL TRIAL: NCT07219862
Title: Evaluating a Clinical Decision Support Tool for Antiretroviral Therapy Optimization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keck School of Medicine of USC (Other)
Collaborators: Los Angeles General Medical Center (Other); AIDS Healthcare Foundation (Other)
Responsible Party: Principal Investigator, Hayoun Lee, Associate Professor, Keck School of Medicine of USC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AI095066
Record Dates: First submitted 2025-10-17; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: HIV (Human Immunodeficiency Virus); Clinical Decision Support System (CDSS); Antiretroviral Therapy, Highly Active; INDIVIDUALIZED THERAPY; AIDS (Acquired Immune Deficiency Syndrome); Personalized Medicine; Precision Medicine
Keywords: hiv; clinical decision support system; antiretroviral therapy; aids; personalized medicine; precision medicine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smART (Experimental): smART (Smart Antiretroviral Therapy Assistant): a digital clinical decision support tool that provides personalized, guideline-based HIV treatment recommendations.
  Interventions: Other: smART (Smart Antiretroviral Therapy Assistant)
- Traditional Prescribing resources (Active Comparator): standard online resources commonly accessed in HIV care, including the Stanford HIV Database, the IAS-USA Drug Resistance Mutations Chart, and the NIH HIV Clinical Guidelines.
  Interventions: Other: Traditional Prescribing resources

INTERVENTIONS:
Other: smART (Smart Antiretroviral Therapy Assistant) — smART is a single-page, offline clinical decision support application that generates personalized HIV treatment recommendations by evaluating over 50,000 possible antiretroviral combinations. The user inputs patient-specific data including genotypic resistance profile, comorbid conditions, drug allergies, concomitant medications, and reproductive status (pregnant or planning pregnancy). smART performs all computations locally and does not store any patient information, ensuring complete data privacy.
  Arms: smART
Other: Traditional Prescribing resources — No additional interventions beyond standard clinical practice will be implemented for study participants. Treatment decisions will be guided by established HIV resources, including the Stanford HIV Database, the IAS-USA Drug Resistance Mutations Chart, and the NIH HIV Clinical Guidelines.
  Arms: Traditional Prescribing resources

SUMMARY:
This study is testing software designed to help healthcare providers choose the best HIV treatment combinations for their patients. HIV medicines, known as antiretroviral therapy (ART), can be complex to manage because the right regimen depends on many factors-such as drug resistance, other health conditions, and medication schedules. Many people with HIV are cared for by general clinicians who may not have access to HIV specialists, which can make treatment decisions more challenging.

In this study, healthcare providers will use patient cases to compare standard HIV treatment resources with a new clinical decision support tool that gives evidence-based ART recommendations at the point of care.

The investigators hypothesize that using the tool will help providers select treatment plans that better match clinical guidelines, make decisions faster, reduce mental effort, and increase overall satisfaction with the prescribing process.

ELIGIBILITY:
Inclusion Criteria:

HIV patients

1. Documented HIV-1 infection
2. Greater than 18 years of age
3. Genotype resistance testing previously conducted or scheduled through clinical care

Providers:

HIV care providers who will determine treatment selections, with or without utilizing our clinical decision support tool

Exclusion Criteria:

HIV patients:

1. Refusal or inability to give informed consent

Providers:

1. Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2028-09-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence of Prescribed ART Regimens to Evidence-Based Recommendations | Assessed at completion of each patient prescribing session at Day 1
  Proportion of antiretroviral therapy (ART) regimens that align with guideline-based recommendations. A regimen is considered adherent if it contains at least three fully active agents (defined as a total drug susceptibility score ≥280) and is not contraindicated based on patient-specific factors identified by the smART tool, including allergies, comorbidities, concomitant medications, pregnancy status, and/or major guideline restrictions.

SECONDARY OUTCOMES:
Proportion of virally suppressed individuals | Assessed at between 1 month and 6 month after completion of each prescribing session
  Viral suppression rates

CONTACTS AND LOCATIONS:
Overall Officials: Hayoun Lee, PhD, Principal Investigator — Keck School of Medicine of USC
Locations (1):
- Los Angeles General Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including drug resistance mutations, comorbidities, comedications, and prescribed regimens, will be shared by publishing manuscripts covering this trial outcomes.
Supporting Information: Study Protocol
Time Frame: The study protocol will be published as supporting information upon completion of the trial and publication of its results.
Access Criteria: Anyone with access to the academic journals publishing this study's results.